CLINICAL TRIAL: NCT07041697
Title: Application of Photobiomodulation Therapy by LED Using a Combined Red and Near-infrared Light Spectrum Improves the Vascular Function of the Radial Artery in Vitro
Brief Title: LED Photobiomodulation Improves Radial Artery Vascular Function in Vitro
Acronym: LED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, André Timóteo Sapalo, Clinical Professor, University of Sao Paulo
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 4.829.712
Record Dates: First submitted 2025-04-25; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Vascular Dysfunction
Keywords: Photobiomodulation; Light-emitting diode; Vascular function; Radial artery

STUDY DESIGN:
Intervention Model Description: To irradiate the arteries, we used a 14 cm × 14 cm LED blanket composed of 30 red-spectrum LEDs (wavelength: 650 nm), delivering a power density of 1.9 mW/cm² and an energy density of 1.7 J/cm² over an irradiation period of 83 seconds. A separate 14 cm × 14 cm infrared LED blanket, also containing 30 LEDs (wavelength: 940 nm), delivered a power density of 1.7 mW/cm² and an energy density of 1.7 J/cm² with an irradiation time of 94 seconds. Additionally, a 14 cm × 14 cm mixed LED blanket, consisting of 18 red (650 nm) and 18 infrared (940 nm) LEDs, provided a power density of 1.7 mW/cm² and an energy density of 0.16 J/cm² over an irradiation period of 73 seconds.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Photobiomodulation Using Red LED Light at 650 nm Wavelength (Experimental): The three arms of the study aim to evaluate the effectiveness of different LED light spectra on vasodilation.
  Interventions: Device: Light-emitting diode photobiomodulation therapy
- Photobiomodulation Using Red LED Light at 940 nm Wavelength (Experimental): The three arms of the study aim to evaluate the effectiveness of different LED light spectra on vasodilation.
  Interventions: Device: Light-emitting diode photobiomodulation therapy
- Photobiomodulation with Combined Red (650 nm) and Infrared (940 nm) LED Light (Experimental): The three arms of the study aim to evaluate the effectiveness of different LED light spectra on vasodilation.
  Interventions: Device: Light-emitting diode photobiomodulation therapy

INTERVENTIONS:
Device: Light-emitting diode photobiomodulation therapy — For the intervention, the isolated arteries were assigned to three experimental groups. The first group (red) was exposed to light at a wavelength of 650 nm for 83 seconds. The second group (infrared) received irradiation at 940 nm for 94 seconds. The third group (mixed) was irradiated with a combination of red (650 nm) and infrared (940 nm) light for 73 seconds.

SUMMARY:
LED photobiomodulation therapy (PBMT) is widely recognized for its beneficial effects in several clinical conditions; however, its potential in modulating vascular function is not yet fully established. Objective: This study aimed to evaluate the application of PBMT by LED (light-emittion diode) using a combined red and near-infrared light spectrum, with a focus on improving the vascular function of the radial artery in vitro. Methodology: A total of 30 radial artery segments were studied and divided into three groups of 10 segments: the PBMT LED group combined with red and infrared light (R + IR), the red light (R) group, and the infrared light (IR) group. Prior to light irradiation at wavelengths of 650 nm and 940 nm, vascular function in these segments was pharmacologically inhibited using L-NAME. The drugs phenylephrine, acetylcholine, and sodium nitroprusside were used to determine if irradiation could restore the inhibited vascular functions. Superoxide anion levels, an important reactive oxygen specie (ROS), were measured using a chemiluminescence assay with lucigenin. The bioavailability of nitric oxide was evaluated using a Griess Reagent Kit assay, while nitric oxide production was assessed through the DAF fluorescence assay. The vascular inflammation was determined by the Intercellular Adhesion Molecule 1 (ICAM-1) expression.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing coronary artery bypass grafting using the radial artery

Exclusion Criteria:

* Patients with poorly compliant radial arteries or those who underwent coronary artery bypass grafting without use of the radial artery were excluded from the study

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-01-12 (Actual); Primary Completion 2024-12-21 (Actual); Study Completion 2025-02-21 (Actual)

PRIMARY OUTCOMES:
Diameter of Isolated Radial Artery Rings (2 mm) | 12 months
  Description of Primary Outcome Measure(s):
  The primary outcome of this study is the evaluation of vascular compliance during vasodilation of isolated radial artery rings (2 mm in diameter), with a specific focus on the effects of LED photobiomodulation on arterial function.

SECONDARY OUTCOMES:
Evaluation of reactive oxygen species (ROS) | 12 months
  Superoxide anion (O₂--) generation, a key reactive oxygen species (ROS), will be measured in arterial tissue from the R + IR, R, and IR groups using a lucigenin-enhanced chemiluminescence assay. Lucigenin will serve as the electron acceptor, and nicotinamide adenine dinucleotide phosphate (NADPH) as the substrate. Results will be expressed as a percentage of concentration.

CONTACTS AND LOCATIONS:
Locations (1):
- University of São Paulo Medical School in Ribeirão Preto, Ribeirão Preto, São Paulo, Brazil

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-22): https://cdn.clinicaltrials.gov/large-docs/97/NCT07041697/Prot_SAP_000.pdf